CLINICAL TRIAL: NCT03296332
Title: Shandong and Ministry of Health Action on Salt and Hypertension Project (SMASH)
Brief Title: Shandong and Ministry of Health Action on Salt and Hypertension Project
Acronym: SMASH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Shandong Province Centers for Disease Control and Prevention (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ma Jixiang, Deputy director, The National Center for Chronic and Noncommunicable Disease Control and Prevetion(NCNCD), Centers for Disease Control and Prevention, China
Other Study IDs: 2012GSF11828
Record Dates: First submitted 2016-05-31; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Hypertension
Keywords: Evaluation; Population-based Intervention; Salt intake; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We used blood samples of 17,160 respondents to test blood glucose and blood lipids and 24-hour urinary samples of 1820 respondents in total to investigate the changes in sodium/salt intake.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This final evaluation intends to evaluate SMASH implementation outcomes and intervention effects through quantitative and qualitative assessment, and provide evidence for the national government to develop salt-reduction and blood-pressure lowering strategies in large scales.

DETAILED DESCRIPTION:
Every year, about 1.65 million people die of excessive salt intake in the world as excessive sodium will raise blood pressure, which further increase prevalence risks of cardiovascular and kidney diseases. Therefore, reducing salt intake has been recognized as one of the most cost-effective measures for health improvement. Adopting critical salt-reduction measures can substantially reduce prevalence risks of cardiovascular and other chronic diseases. In this sense, exploring salt-reduction strategies that are widely effective among populations is critical for prevention and management of cardiovascular diseases.

The daily salt intake currently recommended by WHO is 5g (6g is recommended by Chinese government). It is estimated that 2.50 million people will not die each year if the global salt consumption is lowered to the recommended level. WHO member countries have reached an agreement to reduce 30% of the salt intake of people across the world by 2025. However, there are not enough study evidence and practical foundation for achieving the salt-reduction goal among all human beings.

Shandong is a large Chinese province with 96.85 million permanent population in its 138 counties (districts) and 62,719 communities (villages or municipal neighborhood communities). Shandong has high prevalences of cardiovascular diseases with an adult hypertensive prevalence above the national average. According to the national nutrition survey in 2002, Shandong consumed 12.6g salt per capita for daily cooking, much higher than the recommended amount (6g) in Chinese dietary guidelines. Shandong and the Ministry of Health signed a five-year cooperative agreement in 2011, Shandong-MOH Action on Salt and Hypertension ("SMASH"). The program has adopted multi-angle and multi-level intervention strategies to reduce salt intake by people for the purpose of preventing hypertension and other diseases related to salt.

SMASH baseline survey in 2011 studied 15,350 people aged 18-69 by regions and towns with multi-stage cluster random sampling to investigate their blood pressures and conditions. The survey showed that hypertensive prevalence, awareness, treatment and control rates were 23.4%, 34.5%, 27.5%, 14.9% respectively. In the baseline survey, 24-hour urine of 2,112 people was collected, and a salt intake of 13.8g per person per day was obtained in accordance with the urinary sodium data.

Since the commencement of the program, Shandong provincial government has cooperated with relevant departments to establish a work mechanism that is led by MOH, implemented by professional institutes and extensively engaged by the whole society. The program team has developed food standards and regulations and promoted salt-reduction actions in catering entities, supermarkets and food processing enterprises for a favorable environment of the program. The program team has prepared various publicity materials, and trained key groups (catering workers, food manufacturers, housewives and elementary school students). Salt consumption monitoring points and cardiovascular prevalence monitoring system have been established.

SMASH will conclude in May 2016. In order to assess the intervention course, implementation outcomes and intervention effects, the SMASH program office decided to organize a final evaluation of the program in the whole province in 2016, and quantitative data collection in June and July 2016.

ELIGIBILITY:
Inclusion Criteria:

Permanent residents in the investigated counties (residence more than half a year) at ages between 6 and 69 (ID card ages).

Exclusion Criteria:

1. Residents with severe physical or mental diseases.
2. Urine can't be collected due to aconuresis;
3. The candidate has difficulty to collect urine and can't find an assistant;
4. Patients with acute/chronic urinary tract infection, vaginal infection and perianal infection;
5. Patients with acute hemorrhagic diseases in urinary tract, vagina and digestive tract;
6. Women in pregnancy, lactation and menstrual periods (those whose menstruation finishes for two days are eligible);
7. Patients with severe vomiting and diarrhea symptoms.

Ages: 6 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Respondents are permanent residents in the investigated counties (residence more than half a year) at ages between 6 and 69 (ID card ages), but those with severe physical or mental diseases can't participate. The survey is conducted at the same time as the SMASH baseline survey in June-July 2016. Basic demographic information, disease information, hypertension risk elements, knowledge of salt and hypertension, belief and behavior of respondents will be objectively collected and recorded through questionnaires by trained investigators from respondents. The respondents aged 18-69 are sampled from villages and urban neighborhood communities, while those aged 6-17 are sampled from schools.
Sampling Method: Probability Sample
Enrollment: 17160 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypertension | June-July 2016
  Two blood pressure (BP) measurements were obtained using a standardized mercury sphygmomanometer after a 5-min seated rest and information on history of hypertension was obtained using a standard questionnaire. Hypertension was defined as mean systolic BP (SBP) at least 140 mmHg and/or diastolic BP (DBP) at least 90 mmHg, and/or self-reported current use of antihypertensive medication.
Awareness, treatment, and control of hypertension | June-July 2016
  Caculate the proportion of people reported having hypertension, the proportion of people reported taking medication and the proportion of them had their blood presure controlled (<140/<90 mmHg) among those classified as having hypertension.
Salt intake related awareness, belief and behavior | June-July 2016
  A face to face, close-ended questionnaire was administered by trained public health professionals. Questions collected information on: knowledge, attitudes and practices related to sodium and hypertension (relationship between sodium and hypertension, consequences of hypertension, perception of salt consumption, self-reported consumption, intention to reduce salt consumption, and practices towards reducing sodium consumption). Then caculate the KAP rates.
Salt intake | June-July 2016
  All participants were given written and verbal instructions to collect a 24 h urine sample. The samples were first assayed for creatinine concentration using the picric acid method (ADICON Clinical Laboratory; CAP accredited). The sodium concentration was determined using the direction selective electrode method. Daily salt intake was estimated by assessing 24h urinary sodium excretion based on the assumption that all sodium was ingested in the form of sodium chloride.
Salt sources | June-July 2016
  Determined by respondents filling 72-hour dietary recall questionnaires. Furthermore, the survey team asks district/county salt companies to submit sales volumes of different salt products in 2011-2015 for statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Ma Jixiang, MD, Principal Investigator — The National Center for Chronic and Noncommunicable Disease Control and Prevention(NCNCD)
Locations (1):
- The National Center for Chronic and Noncommunicable Disease Control and Prevention, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang J, Xu AQ, Ma JX, Shi XM, Guo XL, Engelgau M, Yan LX, Li Y, Li YC, Wang HC, Lu ZL, Zhang JY, Liang XF. Dietary sodium intake: knowledge, attitudes and practices in Shandong Province, China, 2011. PLoS One. 2013;8(3):e58973. doi: 10.1371/journal.pone.0058973. Epub 2013 Mar 18. PMID 23527061
- [Result] Bi Z, Liang X, Xu A, Wang L, Shi X, Zhao W, Ma J, Guo X, Zhang X, Zhang J, Ren J, Yan L, Lu Z, Wang H, Tang J, Cai X, Dong J, Zhang J, Chu J, Engelgau M, Yang Q, Hong Y, Wang Y. Hypertension prevalence, awareness, treatment, and control and sodium intake in Shandong Province, China: baseline results from Shandong-Ministry of Health Action on Salt Reduction and Hypertension (SMASH), 2011. Prev Chronic Dis. 2014 May 22;11:E88. doi: 10.5888/pcd11.130423. PMID 24854239
- [Result] Xu J, Wang M, Chen Y, Zhen B, Li J, Luan W, Ning F, Liu H, Ma J, Ma G. Estimation of salt intake by 24-hour urinary sodium excretion: a cross-sectional study in Yantai, China. BMC Public Health. 2014 Feb 8;14:136. doi: 10.1186/1471-2458-14-136. PMID 24507470
- [Result] Zhang JY, Yan LX, Tang JL, Ma JX, Guo XL, Zhao WH, Zhang XF, Li JH, Chu J, Bi ZQ. Estimating daily salt intake based on 24 h urinary sodium excretion in adults aged 18-69 years in Shandong, China. BMJ Open. 2014 Jul 18;4(7):e005089. doi: 10.1136/bmjopen-2014-005089. PMID 25037642
- [Result] Yan L, Ma J, Guo X, Tang J, Zhang J, Lu Z, Wang H, Cai X, Wang L. Urinary albumin excretion and prevalence of microalbuminuria in a general Chinese population: a cross-sectional study. BMC Nephrol. 2014 Oct 13;15:165. doi: 10.1186/1471-2369-15-165. PMID 25308236
- [Result] Li JH, Xu AQ, Lu ZL, Yan LX, Guo XL, Wang HC, Ma JX, Zhang JY, Dong J, Wang LH. Dietary sodium intake and its impact factors in adults of Shandong province. Biomed Environ Sci. 2014 Jul;27(7):564-6. doi: 10.3967/bes2014.087. PMID 25073917
- [Result] Ge Z, Guo X, Chen X, Zhang J, Yan L, Tang J, Cai X, Xu A, Ma J. Are Microalbuminuria and Elevated 24 H Urinary Microalbumin Excretion within Normal Range Associated with Metabolic Syndrome in Chinese Adults? PLoS One. 2015 Sep 17;10(9):e0138410. doi: 10.1371/journal.pone.0138410. eCollection 2015. PMID 26379278
- [Result] Chen X, Guo X, Ma J, Zhang J, Tang J, Yan L, Xu C, Zhang X, Ren J, Lu Z, Zhang G, Dong J, Xu A. Urinary sodium or potassium excretion and blood pressure in adults of Shandong province, China: preliminary results of the SMASH project. J Am Soc Hypertens. 2015 Oct;9(10):754-762. doi: 10.1016/j.jash.2015.07.004. Epub 2015 Jul 26. PMID 26302666 (Retraction: PMID 27155247 J Am Soc Hypertens. 2016 May;10(5):472)
- [Result] Ge Z, Zhang J, Chen X, Yan L, Guo X, Lu Z, Xu A, Ma J. Are 24 h urinary sodium excretion and sodium:potassium independently associated with obesity in Chinese adults? Public Health Nutr. 2016 Apr;19(6):1074-80. doi: 10.1017/S136898001500230X. Epub 2015 Jul 31. PMID 26228639
- [Result] Yan L, Bi Z, Tang J, Wang L, Yang Q, Guo X, Cogswell ME, Zhang X, Hong Y, Engelgau M, Zhang J, Elliott P, Angell SY, Ma J. Relationships Between Blood Pressure and 24-Hour Urinary Excretion of Sodium and Potassium by Body Mass Index Status in Chinese Adults. J Clin Hypertens (Greenwich). 2015 Dec;17(12):916-25. doi: 10.1111/jch.12658. Epub 2015 Aug 29. PMID 26332433
- [Result] Zhang J, Guo XL, Seo DC, Xu AQ, Xun PC, Ma JX, Shi XM, Li N, Yan LX, Li Y, Lu ZL, Zhang JY, Tang JL, Ren J, Zhao WH, Liang XF. Inaccuracy of Self-reported Low Sodium Diet among Chinese: Findings from Baseline Survey for Shandong & Ministry of Health Action on Salt and Hypertension (SMASH) Project. Biomed Environ Sci. 2015 Feb;28(2):161-7. doi: 10.3967/bes2015.022. PMID 25716570